CLINICAL TRIAL: NCT06501235
Title: Barriers vs. Resources: A Mechanistic Randomized Clinical Trial Comparing Virtue-Based and Cognitive-Behavioral Interventions in Patients With Chronic Medical Disease
Brief Title: Virtue-Based vs. Cognitive-Behavioral Interventions in Patients With Chronic Medical Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Ausias Cebolla, Assistant Professor of Psychology, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEB-MAR-2023-01
Record Dates: First submitted 2024-06-28; First posted 2024-07-15 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Well-Being, Psychological
Keywords: well-being; cognitive-behavioral intervention; virtue-based intervention
MeSH Terms: conditions — Psychological Well-Being | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Between subjects design
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive-Behavioral Therapy (CBT) (Experimental): This group will receive a 9-week CBT intervention.
  Interventions: Behavioral: Cognitive-Behavioral Therapy (CBT)
- Virtue-Based Intervention (VBI) (Experimental): This group will receive a 9-week VBI intervention.
  Interventions: Behavioral: Virtue-Based Intervention (VBI)

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy (CBT) — An adaptation of the Robles and Peralta's (2010) stress management program will be followed. This program includes key techniques from the CBT approach, such as deactivation techniques, cognitive restructuring, and assertiveness training.
  Arms: Cognitive-Behavioral Therapy (CBT)
Behavioral: Virtue-Based Intervention (VBI) — A Well-being Training based on Contemplative Practices (WTCP) (Cebolla & Alvear, 2019; Alvear & Cebolla, 2023) will be followed. WTCP combines mindfulness practices with various activities based on virtues such as gratitude, altruism, or compassion. This program focuses on generative or constructive meditations, and puts special emphasis on virtuous actions, emotion regulation (both positive and negative emotions) and compassion, and includes strategies from positive psychology, such as strengths-based interventions, savoring, kindness, or the three good things.
  Arms: Virtue-Based Intervention (VBI)

SUMMARY:
The aim of this study is to analyze the specific and common mechanisms of change of two active treatments, one based on reducing barriers -Cognitive Behavioral Therapy (CBT)- and the other based on enhance resources -Virtue-Based Intervention (VBI)- for increasing well-being in patients with chronic medical disease. A mechanistic randomized controlled trial will be conducted with two experimental conditions (CBT and VBI) and four evaluation points (pre- and post-intervention and 6- and 12-month follow-up).

DETAILED DESCRIPTION:
Currently, there are several effective interventions to increase well-being, such as Cognitive-Behavioral Therapy (CBT), which focuses on reducing deficits, and Virtue-Based Interventions (VBI), which focus on encouraging actions that promote well-being. However, there is little research on the mechanisms by which these interventions work. The aim of this study is to analyze the specific and common mechanisms of change of two active treatments (CBT and VBI) for increasing well-being in patients with chronic diseases. This population will be used because of their low level of well-being compared to the general population. A randomized controlled trial will be conducted, with two experimental conditions (VBI and CBT) and four assessment points (pre- and post-intervention, and 6- and 12-month follow-up). We will primarily assess well-being, anxiety, depression, mechanisms specific to each intervention (e.g., dysfunctional thoughts in CBT, use of strengths in VBI), and mechanisms common to psychological interventions (e.g., trust in treatment). First, participants will be screened for eligibility according to the inclusion/exclusion criteria. Second, eligible participants will be randomized to a CBT or VBI condition and will complete baseline measures. Third, participants will receive the core intervention for 9 weeks. Finally, participants will complete measures after treatment and 6 and 12 months later. During treatment, they will answer some questions daily to assess well-being and well-being competencies using Ecological Momentary Assessment (EMA). The hypotheses are: (1) both participants in the CBT and VBI conditions will increase their levels of well-being and the changes will be mediated by the specific mechanisms of each intervention, (2) some of the changes in well-being that may exist in both interventions will be explained by the common factors, (3) all of these changes will be moderated by baseline levels of anxiety, depression and well-being, and (4) both participants in the CBT and VBI conditions will reduce levels of anxiety and depression. The study will be conducted following the principles stated in the Declaration of Helsinki.

Analysis plan:

A mixed approach between quantitative and qualitative methods was applied. Regarding the quantitative methods, differences between groups in demographics and other clinical variables will be tested with T-tests for continuous variables and χ2 tests for categorical variables. Assumptions will be tested and, if broken, non-parametric and robust alternatives will be applied. Relations between continuous variables will be screened and tested for differences between groups. In addition, reliability of self-report variables will be assessed to ensure good psychometric properties.

To test the impact of VBI and CBT across time, a two-way mixed Analysis of Covariance (ANCOVAs) will be implemented (group as between-subjects variable, time as a within-subjects variable). Main and interaction effects will be estimated, along with post hoc tests with correction of type I errors (Bonferroni and Šidák) and estimated marginal means with 95% confidence intervals. Assumptions for ANCOVA will be tested and corrections will be implemented if broken. All contrasts will count with effect sizes and 95% confidence intervals. Dropout and other missing data patterns will be assessed. More concretely, proportion of missing data will be screened and compared across groups. If relevant or non-ignorable missingness is found, multiple imputation of missing data will be applied. More concretely, a multilevel strategy will be implemented. Predictors will be selected by design and by sharing a relevant amount of variance with each outcome. In addition, sensitivity analysis will be implemented to test robustness of imputation models. To estimate the impact of sample size, all analysis will count with a sensitivity analysis will be implemented at 90% power and 95% confidence using G*Power 3.1.

To analyze potential mechanisms of change in each program, structural equation models (SEM) will be implemented. Difference scores between times (post - pre intervention and follow ups - pre intervention) will be computed and implemented as outcomes. Following our framework, a series of proposals of mechanisms will be developed as theoretical models for the SEM. Given most or all variables will be continuous, Maximum Likelihood Robust will be used as the estimation method along with robust standard errors of estimates (this enables unbiasing estimates from deviations from normality). Missing data will be handled with the Full-Information Maximum Likelihood method. Fit will be assessed with indices and thresholds recommended by literature. Due to mediations present in our framework, indirect effects will be estimated with bootstrap techniques. In addition, a correction for multiple testing will be applied due to the proposal of several theoretical models. A power analysis revealed with 90% power, 95% confidence, and 210 degrees of freedom (20 variables), a minimum sample size of n = 100 able to differentiate between a population RMSEA = 0.5 with an alternative RMSEA = 0.08. However, sample size will be increased if available.

To analyze the EMA scores, multilevel longitudinal models will be implemented. More concretely, the specific time of assessment nested in the overall times (pre, post, and follow-ups), nested in individuals, and then nested in groups (VBI or CBT). Available models will be screened (e.g., cross-lagged growth modelling, GIMME models, dynamic SEM) and employed.

Descriptives, bivariate tests, and ANCOVAs will be estimated with JASP, while SEM and EMA analyses will be estimated with the R environment. Specific packages are lavaan, lme4 y EMAtools.

Regarding the qualitative methods, semi-structured interviews will be implemented with an inductive perspective to search for underlying categories to participants responses. Thematic analysis will be used as framework to locate and describe these categories. Two members of the team will develop the thematic analysis with the following phases: (1) reading and re-reading of open-ended responses and describe general ideas; (2) generation of first codes by extracting all relevant verbal information regarding research questions, assigning a brief description or code, and allocating them in a table; (3) organizing the codes in the search of themes; (4) review the proposed themes aiming for homogeneity and specificity of contents, and ensuring units of verbal meaning are adequately represented in the themes; (5) definition and description of themes.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 70 years old.
2. Able to read and write in Spanish.
3. Having a computer with internet access in a safe place (home or private office) and the skills to use it.
4. Having a low level of well-being (i.e., a score of less than 13 on the WHO well-being index, assessed with the WHO-5 questionnaire).
5. Having a diagnosis of a chronic medical disease (diabetes, epilepsy, cancer, etc.) according to standard criteria.

Exclusion Criteria:

1. Diagnosis of a mental disorder assessed with the Spanish edition of the Mini-International Neuropsychiatric Interview (MINI).
2. Complications of the chronic medical disease that require hospital treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mental Health Continuum Scale (MHC-SF; Keyes, 2009) | Before (week 0) and after (week 9) intervention
  This 14-item scale measures emotional, social, and psychological well-being. It assesses the frequency of feeling a certain way during the last month. The Spanish version of Echevarría et al. (2017) will be used.
Cognitive Therapy Scale-Self Report (CCTS-SR) (Strunk et al., 2014) | Before (week 0) and after (week 9) intervention
  This 29-item scale measures the use of CBT skills during the last 2 weeks. The scale will be translated and adapted for use in this study.
Well-being Competencies Scale (WCS) | Before (week 0) and after (week 9) intervention
  This 16-item ad hoc scale was constructed to assess several well-being skills (e.g., mindfulness, savoring, gratitude) that are trained in the Well-being Training Based on Contemplative Practices (WTCP).
Generic Sense of Ability to Adapt Scale (GSAAS; Franken et al., 2023) | Before (week 0) and after (week 9) intervention
  This 10-item scale measures the ability to readjust after a personally challenging event (e.g., "I can handle setbacks well"). The scale will be translated and adapted for use in this study.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder Questionnaire (GAD-7; Spitzer et al., 2006) | Before (week 0) and after (week 9) intervention
  This 7-item instrument measures the presence of anxious symptoms in the last 15 days. Higher scores indicate a greater presence of anxious symptomatology. The Spanish version of García-Campayo et al. (2010) will be used.
Patient Health Questionnaire-9 (PHQ-9; Kroenke et al., 2001) | Before (week 0) and after (week 9) intervention
  This 9-item instrument measures the presence of depressive symptoms in the last 2 weeks. The severity of symptomatology is classified into 4 levels: 0-4 (minimal), 5-9 (mild), 10-14 (moderate), 15-19 (moderate-severe), and 20-27 (severe). The Spanish version of Diez-Quevedo et al. (2001) will be used.
Well-Being Locus of Control Scale (WB-LOC12; Farier et al., 2021) | Before (week 0) and after (week 9) intervention
  This 12-item scale measures the degree of expectancy about well-being control. It is composed of three factors: internal, others, and opportunities. The scale will be translated and adapted for use in this study.
Compassion Motivation and Action Scales (CMAS; Steindl et al., 2021) | Before (week 0) and after (week 9) intervention
  This instrument encompasses two dimensions assessing self-compassion and compassion to others' motivation and action. The self-compassion dimension encompasses 18 items, and the compassion to others dimension includes 12 items. The scale will be translated and adapted for use in this study.
Therapeutic Factors Inventory-Short Form (TFI-S; MacNair-Semands et al., 2010) | After session 4 (week 4) and after (week 9) intervention
  Compassion Motivation and Action Scales (CMAS; Steindl et al., 2021)
MPOQ-Common Factor Scale (Finsrud et al., 2021) | After session 4 (week 4) and after (week 9) intervention
  This 14-item scale assesses common relational factors in psychological treatments. It includes two factors: trust in the therapist and trust in the treatment. The scale will be translated and adapted for use in this study.
Diabetes Distress Scale (DDS; Polonsky et al., 2005) | Before (week 0) and after (week 9) intervention
  This 17-item instrument measures stress symptoms related to suffering from diabetes in the last month. It includes 4 factors: emotional stress, physician stress, regimen stress, and interpersonal stress. The Spanish version of Ortiz et al. (2013) will be used.
Quality of life in epilepsy-31 inventory (QOLIE-31-P; Cramer et al., 1998) | Before (week 0) and after (week 9) intervention
  This 39-item instrument assesses quality of life of patients with epilepsy, including 7 factors: energy/fatigue, mood, daily activities, cognition, medication effects, seizure worry, and overall quality of life. The Spanish version of Sarudiansky et al. (2023) will be used.

OTHER OUTCOMES:
WHO-5 Questionnaire | Before intervention (screening)
  The World Health Organization's 5-item Well-Being Index (WHO-5) is a brief, generic global rating scale that measures subjective well-being. It assesses how often participants felt a certain way during the past two weeks.
MINI International Neuropsychiatric Interview (MINI) 5.0 | Before intervention (screening)
  This is a structured diagnostic psychiatric interview used by mental health professionals to assess a range of psychiatric disorders according to the Diagnostic and Statistical Manual of Mental Disorders and the International Classification of Diseases. It's a standardized tool used in clinical and research settings to help diagnose conditions such as depression, anxiety disorders, and bipolar disorder.
Sociodemographic variables | Before intervention (screening)
  Information on sex, gender, marital status, educational level, and employment status, will be collected.
Adherence | After (week 9) intervention
  It will be evaluated through the presence of the sessions and completion of homework assignments.
Satisfaction and opinion with intervention | After (week 9) intervention
  Ad hoc questions will be asked about satisfaction and opinion about the treatment.
Ecological Momentary Assessment | Daily, from one week before the start of the intervention until one week after the end of the intervention (i.e., during 70 days).
  The level of well-being and the competencies from the Wellbeing Training based on Contemplative Practices (WTCP) were assessed daily using the m-Path app (https://m-path.io/landing/) with nine ad hoc items.

CONTACTS AND LOCATIONS:
Overall Officials: Ausiàs Cebolla Martí, PhD, Principal Investigator — Univeristy of Valencia
Locations (1):
- Faculty of Psychology and Speech Therapy, University of Valencia Valencia, Comunidad Valenciana, Spain, 46010, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Upload databases to OSF (https://osf.io/)
Supporting Information: SAP, Analytic Code
Time Frame: Following the publication of the article
Access Criteria: Open access

REFERENCES:
- [Background] Alvear, D., & Cebolla, A. (2023). La ciencia de la virtud. Manual de Entrenamiento en Bienestar basado en prácticas Contemplativas (EBC). Kairós. Cebolla, A., Herrero, R., Carrillo, A., Navarro, J., Soler, J., & Alvear, D. (2019). Contemplative practice-based well-being training (CBWT): Towards a contemplative positive psychology. In L. Galiana & N. Sansó (Eds.), The power of compassion (pp. 159-174). Nova Science Publishers. Keyes, C. L. M. (2009). Atlanta: Brief description of the mental health continuum short form (MHC-SF). Retrieved from https://peplab.web.unc.edu/wp-content/uploads/sites/18901/2018/11/MHC-SFoverview.pdf Robles, H., & Peralta, M. I. (2010). Programa para el control del estrés. Pirámide. Sarudiansky, M., Lanzillotti, A. I., Gerbaudo, M. A., Wolfzun, C., Kochen, S., Stivala, E., d'Alessio, L., & Korman, G. P. (2023). Cultural adaptation and psychometric properties of the Patient-weighted Quality of Life in Epilepsy 31 Inventory (QOLIE-31P) in Argentina. Epilepsy & Behavior, 141, 109132. https://doi.org/10.1016/j.yebeh.2023.109132